CLINICAL TRIAL: NCT04724057
Title: Post Marketing Clinical Trial to Demonstrate the Performance of the MedHub AutocathFFR Device.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medhub Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLN-FFR-002
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease
Keywords: AutocathFFR; Medhub; FFR
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: AutocathFFR — The MedHub Autocath FFR device is a software only medical device. The FFR is computed from several standard DICOM format 2D angiography images retrieved from the C-arm imaging system, which display the structure of the vessels. The MedHub AutocathFFR device software analyzes these images and automatically (without the need for user selection or markings) and computes and displays the FFR on the viewed blood vessel.

SUMMARY:
Patients with suspected coronary artery disease who are scheduled to undergo a coronary angiography procedure will be enrolled in the study. The angiographic images will be processed by the Medhub Autocath FFR device to generate the Autocath FFR measurement. Based on AMAR approval, MedHub Autocath FFR measurements may be used to determine revascularization in lesions found in the Left Anterior Descending (LAD) coronary artery. Consequently, invasive FFR (using a coronary pressure wire and hyperemic stimulus) is not mandatory for lesions in the LAD, although it is at the discretion of the physician whether or not to perform the invasive FFR procedure. Lesions in the Right Coronary Artery (RCA) and Left Circumflex Coronary (LCX) arteries, when clinically indicated, will be required to undergo an invasive FFR procedure in order to determine revascularization. In these cases, the Autocath FFR measurements will not be used for diagnostic or clinical decisions, but solely as a supportive tool. The MedHub Autocath FFR measurement per vessel will be compared to the invasive FFR measurement in the RCA and LCX lesions and in LAD lesions, for which invasive FFR measurements are available.

The dichotomously scored MedHub Autocath FFR per vessel will be compared to the invasive FFR, where an FFR ≤ 0.80 will be considered "positive", while an FFR > 0.8 will be considered "negative". The sensitivity and specificity of the MedHub Autocath FFR will be calculated.

DETAILED DESCRIPTION:
The proposed study is designed to assess performance and safety data for the MedHub Autocath FFR device.

The study is a prospective, multi-center, single-arm, post-marketing study. A total of 488 subjects will be enrolled in the study. The study population who represent the target population for this procedure consists of subjects with known or suspected coronary artery disease (CAD) who are scheduled to undergo a coronary angiography procedure and on whom invasive FFR will be measured in vessels with meaningful coronary lesions. Patients of both genders, all ethnicities, >18 years of age will be recruited to the study. Study subjects will be enrolled from numerous hospitals in Israel.

Investigators will screen subjects based on the inclusion/exclusion criteria described below. General patient demographics, medical history, concomitant medications, C-arm angiography system used, FFR pressure wire used, etc., will be obtained for study subject.

Subjects with known or suspected coronary artery disease who are scheduled for clinically indicated invasive coronary angiography will comprise the patient population. Coronary angiography will be performed in a routine fashion in patients with suspected coronary artery disease. The collected diagnostic angiography images will be processed using the Medhub Autocath FFR device to generate the Autocath FFR. Based on operator's discretion, the location of the stenosis and when clinically indicated, invasive FFR will be measured using a coronary pressure wire and hyperemic stimulus.

The patient's angiographic images will be processed using the MedHub Autocath FFR device. Based on AMAR approval, MedHub Autocath FFR measurements may be used to determine revascularization in lesions found in the Left Anterior Descending (LAD) coronary artery. Consequently, invasive FFR will not be mandatory for lesions in the LAD, and it will be at the discretion of the physician whether or not to perform the invasive FFR procedure. Lesions in the Right Coronary Anterior (RCA) and Left Circumflex (LCX) arteries, when clinically indicated, will be required to undergo an invasive FFR procedure in order to determine revascularization. That is, in these cases the MedHub Autocath FFR measurements will not be used for diagnostic or clinical decisions, but solely as a supportive tool. The MedHub Autocath FFR measurement per vessel will be compared to the invasive FFR measurement in the RCA and LCX lesions and in LAD lesions, for which invasive FFR measurements are available.

The dichotomously scored MedHub Autocath FFR per vessel will be compared to the invasive FFR, where an FFR ≤ 0.80 will be considered "positive", while an FFR > 0.8 will be considered "negative". The sensitivity and specificity of the MedHub Autocath FFR will be calculated. Furthermore, the MedHub Autocath FFR accuracy, positive predictive value and negative predictive value per vessel and per lesion will be determined.

Usability of the MedHub Autocath FFR device will also be assessed including User Manual comprehension and usability of the device in the hands of the users (i.e., interventional cardiologists).

Details on the timing of all study procedures are given in the Time and Events Schedule in Attachment B of the Protocol. The anticipated enrollment period is approximately 6 months and therefore, the complete duration of the study is expected to last 8-9 months, during which time 488 patients will be enrolled at 3-5 sites.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Subjects with suspected coronary artery disease who are scheduled to undergo a coronary angiography procedure.
* Subject is planned to undergo an invasive FFR with IV or intracoronary Adenosine, Adenosine Triphosphate (ATP) or Papaverine used as hyperemic stimulus*.

  * Not mandatory for lesions in the LAD

Exclusion Criteria:

* Vessel size less than 2 mm.
* CTO in target vessel.
* Prior CABG, heart transplant or valve surgery, prior TAVI/TAVR or severe left sided valvular disease.
* TIMI Grade 2 or lower.
* Target lesion involves Left Main (stenosis >50%).
* Severe, diffuse disease defined as the presence of diffuse, serial gross luminal irregularities present in the majority of the coronary tree.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity | Immediate after procedure
  Co-primary endpoints are the sensitivity and specificity of the dichotomously scored MedHub Autocath FFR per vessel compared to invasive FFR, where an FFR ≤ 0.80 is scored "positive", while an FFR > 0.8 is considered "negative".